CLINICAL TRIAL: NCT02474095
Title: Two Versus Four Times-Weekly ALTENS for Treatment of Radiation-Induced Xerostomia: A Pilot Study
Brief Title: Acupuncture-Like Transcutaneous Electrical Nerve Stimulation in Treating Radiation-Induced Xerostomia in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 247213; NCI-2015-00823 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 247213 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Carcinoma; Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (ALTENS QIW) (Experimental): Patients undergo ALTENS delivered via the Codetron machine QIW for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Transcutaneous Acupoint Electrical Stimulation
- Arm II (ALTENS BIW) (Active Comparator): Patients undergo ALTENS delivered via the Codetron machine BIW for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Transcutaneous Acupoint Electrical Stimulation

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Transcutaneous Acupoint Electrical Stimulation — Undergo ALTENS
  Other Names: acupuncture-like transcutaneous electrical nerve stimulation; ALTENS; TAES

SUMMARY:
This randomized pilot clinical trial studies alternate schedules for acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) in treating dry mouth (xerostomia) caused by radiation therapy (RT) in patients with head and neck cancer. ALTENS is a procedure in which mild electric currents are applied to certain acupuncture points on the body and may help relieve dry mouth caused by RT and improve quality of life. It is not yet known whether giving ALTENS more frequently works better than standard ALTENS in treating dry mouth caused by RT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether ALTENS treatment using a four-times weekly schedule for 6 weeks reduces overall xerostomia burden, using the University of Michigan 15-item Xerostomia-related Quality of Life Scale (XeQoLS), compared to the standard ALTENAS schedule of twice-weekly for 12 weeks, at 15 months from the start of ALTENS treatment.

SECONDARY OBJECTIVES:

I. Determine whether ALTENS treatment using a four-times weekly schedule for 6 weeks reduces overall xerostomia burden, using the University of Michigan 15-item Xerostomia-related Quality of Life Scale (XeQoLS), compared to the standard ALTENS schedule of twice-weekly for 12 weeks, at 6, 9, 15, and 21 months from the start of ALTENS treatment.

II. Examine the benefit of ALTENS treatment using a four-times weekly schedule for 6 weeks on overall quality of life, using the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire, QLQ-C30, including the questionnaire module specific to head and neck cancers (QLQ-H&N35), compared to the standard ALTENS schedule of twice-weekly for 12 weeks, at 6, 9, 15, and 21 months from the start of ALTENS treatment.

III. To compare the toxicity between treatment schedules using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE Version 4.0).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo ALTENS delivered via the Codetron machine four times weekly (QIW) for 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo ALTENS delivered via the Codetron machine twice-weekly (BIW) for 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6, 9, 15, and 21 months.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Must have received and completed radiotherapy with or without chemotherapy for head and neck cancer; time from completion of radiotherapy to registration must be at least 3 months and up to a maximum of 1 year
* Have grade 1 or 2 symptomatic dry mouth (xerostomia) according to CTEP NCI Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
* Have complete history and physical examination documenting no clinical evidence of disease within 8 weeks of registration
* After completion of radiotherapy, within the last 12 months, a positron emission tomography (PET)/computed tomography (CT) or contrast-enhanced CT scan must be performed within 8 weeks of registration demonstrating no evidence of disease or loco-regional recurrence
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with normal saliva production (no salivary gland changes; no xerostomia)
* Patients who are on pilocarpine for ophthalmic or non-ophthalmic indications
* Patients who are on regular medications which will induce xerostomia (tricyclic antidepressants, antihistamines with anticholinergic effects)
* Patients with Sjogren's syndrome
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive ALTENS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Change in XeQoLS | Baseline to 15 months
  A repeated measures model will be used to compare XeQoLS scores between the two arms at 15 months. Additional analysis will be performed using an area-under-the-curve (AUC) comparison of XeQoLS functional scores and the EORTC QLQ-C30 and the EORTC-QLQ-H&N35 scores between the two groups over time.

SECONDARY OUTCOMES:
Change in the quality of life using the EORTC QLQ-C30 and the EORTC-QLQ-H&N35 | Baseline to up to 21 months
  A repeated measures model will be used to compare EORTC QLQ-C30 and the EORTC-QLQ-H&N35 scores between the two arms. Additional analysis will be performed using an AUC comparison of XeQoLS functional scores and the EORTC QLQ-C30 and the EORTC-QLQ-H&N35 scores between the two groups over time.
Change in XeQoLS | Baseline to up to 21 months
  A repeated measures model will be used to compare XeQoLS scores between the two arms. Additional analysis will be performed using an AUC comparison of XeQoLS functional scores and the EORTC QLQ-C30 and the EORTC-QLQ-H&N35 scores between the two groups over time.
Incidence of adverse events between treatment schedules using CTEP NCI CTCAE version 4.0 | Up to 30 days after the last intervention or a new treatment is started
  The frequency of toxicities will be tabulated by grade.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States